CLINICAL TRIAL: NCT03692520
Title: Recombinant Anti-EGFR Monoclonal Antibody（SCT200）in Patients With Advanced Solid Tumors or Lymphoma : A Phase Ⅰb, Open-label, Multicenter Study.
Brief Title: Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of SCT200 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT200-X101
Record Dates: First submitted 2018-09-29; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-06

CONDITIONS: Advanced Solid Tumors
Keywords: Neoplasms; Solid Tumors; Epidermal growth factor receptor; EGFR; SCT200
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCT200 (Experimental): Initially, SCT200 6.0mg/kg will be administered at day 1 every week for a maximum of 6 cycles. After 6 cycles SCT200 8.0mg/kg will be administered at day 2 every weeks until disease progression
  Interventions: Biological: SCT200

INTERVENTIONS:
Biological: SCT200 — Recombinant Anti-EGFR Monoclonal Antibody （SCT200）

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of recombinant anti-EGFR monoclonal antibody（SCT200）in patients with advanced solid tumors treated after failure of standard therapy.

DETAILED DESCRIPTION:
This open label, multicenter phase Ib study is designed to evaluate Objective Response Rate (ORR) in advanced solid tumors (gastric/gastroesophageal junction cancer, hepatocellular carcinoma,pancreatic cancer,gallbladder cancer/bile duct cancer，renal cell carcinoma，ovarian cancer，or other advanced solid tumor) treated with anti-EGFR monoclonal antibody SCT200.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and can understand and comply with the requirements of the study;
* Males or females. Aged 18 to 75 years old;
* Life expectancy of longer than 3 months ( clinical assessment);
* With an Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
* Histological or cytological diagnosis of advanced solid tumors(gastric/gastroesophageal junction cancer, hepatocellular carcinoma,pancreatic cancer,gallbladder cancer/bile duct cancer，renal cell carcinoma，ovarian cancer，other advanced solid tumor)
* Advanced solid tumor or lymphoma wuth failure of standard treatment;
* According to RECIST 1.1 , patients must have at least one measurable lesion that can be accurately assessed;
* Adequate organ and marrow function as defined below:

Absolute neutrophil count (ANC) greater than/equal to 1.5×l09/L; Platelets greater than/equal to 75×109/L; Hemoglobin greater than/equal to 80g/L; Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than/equal to 3 times ULN, or less than/equal to 5 times ULN if known liver metastases; Total bilirubin less than/equal to 1.5 within institutional limit of normal (ULN); Serum creatinine less than/equal to 1.5 times ULN; Electrolyte: magnesium greater than/equal to normal.

Exclusion Criteria:

* Patients who are allergic to analogue of SCT200 and/or its inactive ingredients;
* Patients with active central nervous system metastasis or a history of central nervous system metastasis;(If the subject has been suspected with central nervous system metastasis,imaging examination confirmation must be performed within 28 days to exclude central nervous system metastasis;
* Subject receiving bisphosphonate or denosumab treatment for bone metastases was initiated within 28 days prior to study. (If the subject has received bisphosphonate or denosumab treatment prior to study and showing stable time at least 28 days,the subject will be allowed to use it.) Subjects who were enrolled in this study may start taking bisphosphonate or denosumab for bone metastases after the first assessment of the efficacy.
* Patients with other primary malignancies, except cured of basal cell carcinoma skin cancer, carcinoma in situ of cervix, or prostatic intraepithelial neoplasia;
* Patients administrated EGFR target treatment including EGFR TKI agent or anti- EGFR monoclonal antibody;
* Within 4 weeks, patients received anti-tumor drugs (such as chemotherapy, hormone therapy, immune therapy, the antibody therapy, radiotherapy) or research drugs, or patients with grade 2 or more adverse reaction caused by previous anti-tumor therapy(except alopecia or neurotoxicity grade 2 or less);
* Patients are currently enrolled in other research devices or in research drugs, or less than 4 weeks from other research drugs or devices.
* Prior to the first dose of study drug, patients received major surgery requiring general anesthesia has been completed less than 4 weeks; surgery requiring local anesthesia/epidural anesthesia has been completed less than 72 hours; skin biopsy requiring local anesthesia has been completed less than 1 hour.
* Patients treated with EPO, G-CSF or GM-CSF.
* Patients who have clinically significant cardiovascular disease (defined as unstable angina pectoris, symptomatic congestive heart failure (NYHA, greater than II), uncontrollable severe arrhythmia);
* Patients occurred myocardial infarction within 6 months.
* Patients who have interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, or CT or MRI reminder ILD .
* Patients with clinical symptoms, required clinical intervention or stable time less than 4 weeks of serous cavity effusion (such as pleural effusion and ascites);
* Patients with medical or psychiatric condition or laboratory abnormality may interfere with the interpretation of study results;
* Pregnant or lactating women, or women who planned to be pregnant within 6 months of treatment;
* Patients who were not willing to accept effective contraceptive measures (including male or female subjects) during treatment and for at least 6 months after your last dose of SCT200;
* Patients with active hepatitis B or active hepatitis C, etc. (for patients with a history of hepatitis B, whether treated or not, HBV DNA ≥104 or ≥ 2000IU/ml, HCV RNA≥15IU/ml); HIV antibody positive (if there is no clinical evidence suggesting HIV infection, there is no need to detect);
* Patients with uncontrolled active infections within 2 weeks before enrollment (except urinary tract infection or upper respiratory tract infection);
* Patients have alcohol or drug addiction;
* Subjects who are considered unsuitable for participating in this study for various reasons at the discretion of the investigator，such as inability to comply with study and/or follow-up procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-09-30 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 year
  ORR is defined as proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 during trial treatment.

SECONDARY OUTCOMES:
Adverse events (AEs) | 1 year
  AE are assessed according to NCI CTCAE v4.03.
Progress Free Survival ( PFS) | 1 year
  PFS is defined as the time from first dose of SCT200 until the date of first documentation of progression or date of death, whichever occurs first,according to RECIST v1.1 criteria.
Disease control rate (DCR) | 1 year
  The achievement of any a stable response（SD）, partial response (PR) or complete response (CR), according to RECIST v1.1 criteria.
Overall survival (OS) | 1 year
  OS is defined as time from first dose of SCT200 until the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: jianming xu, MD, Principal Investigator — 307 Hospital of PLA
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No